CLINICAL TRIAL: NCT03603119
Title: A Comparison of Midazolam Versus Dexamethasone-ondansetron in Preventing Postoperative Nausea-vomiting in High Risk Patients Undergoing Laparoscopic Surgeries
Brief Title: Midazolam Versus Dexamethasone-ondansetron in Preventing Postoperative Nausea-vomiting for Laparoscopic Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PONV prophylaxis
Record Dates: First submitted 2018-06-02; First posted 2018-07-27 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting; Dexamethasone; Ondansetron; Midazolam; Laparoscopy; High risk
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Saline Solution; Midazolam; Dexamethasone; Ondansetron

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: concealed envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Dexamethasone-ondansetron
  Interventions: Drug: Dexamethasone, ondansetron
- Group B (Experimental): Midazolam
  Interventions: Drug: Normal saline, Midazolam

INTERVENTIONS:
Drug: Normal saline, Midazolam — 2 cc normal saline i.v. after anaesthesia induction.2 mg of injection midazolam intravenous 30 minutes prior to the end of surgery
  Arms: Group B
Drug: Dexamethasone, ondansetron — 8mg of dexamethasone i.v. after anaesthesia induction and 4 mg of ondansetron i.v. 30 minutes prior to the end of surgery.
  Arms: Group A

SUMMARY:
Postoperative nausea and vomiting(PONV) affects 11 to 60 % of patients undergoing surgery and is a major cause of postoperative morbidity. Risk factors include female gender, non smokers, postoperative use of opioids and a past history of PONV. The simplified Apfel risk score is used to identify patients at risk for PONV. PONV prophylaxis is provided intraoperatively to patients with 2 or more risk factors. In spite of numerous drugs available, control of PONV remains a difficult task. Midazolam is a commonly used drug perioperatively for its anxiolytic and sedative properties. It decreases analgesic requirement and has also been found to have an antiemetic effect. This present study is designed to compare the prophylactic use of iv midazolam with a commonly used combination of dexamethasone-ondansetron in high risk patients (as defined by the modified Apfel score) undergoing laparoscopic surgeries.

DETAILED DESCRIPTION:
After Institutional Ethical Committee approval and written informed consent, 120 adult patients will be recruited for the study if they satisfy the inclusion and exclusion criteria as mentioned later. Consent will be obtained from the patients themselves. Standard protocol for administration of anaesthesia will be followed in all patients which is briefly described. All patients will receive general anaesthesia and will be induced with Propofol titrated to effect. Intraoperatively, isoflurane will be used as maintenance agent and vecuronium or atracurium as non depolarizing muscle relaxant. For analgesia, patients will receive intraoperative fentanyl.

For the purpose of the study, patients will be randomized into two groups depending upon a computer generated randomized sheet. Group A will receive 8mg of dexamethasone i.v. after anaesthesia induction and 4 mg of ondansetron i.v. 30 minutes prior to the end of surgery. Patients in Group B will be administered 2 mg of midazolam i.v. 30 minutes prior to the end of surgery. Time to achieve Post anaesthesia discharge score( PADSS) of ≥9 will be noted. Patients will be asked to report any incidence of nausea, retching or vomiting for the first 24 hours after surgery. The incidence of PONV and the amount of rescue antiemetic received will be noted at 2 hours and at 24 hours postoperatively. PONV will be scored based on the PONV Impact Scale score questionnaire (mentioned in the proforma)12. Rescue antiemetics will be administered in case the patient complains of PONV in accordance with American society of anesthesiologists (ASA) guidelines. The first line of rescue in Group A will be 10 mg of iv metaclopromide. Antihistaminics will be the second line of rescue antiemetic. In group B the first line of antiemetic will be 4 mg of ondansetron i.v. 10 mg of iv metaclopromide will be second line of rescue drug.

Study period : It is estimated that the study will be completed within one year Sample size Assuming a reduction in 45 % in the incidence of PONV, with α error of 0.05 and β of 0.02, we would require 60 patients in each group i.e. a total of 120 patients.13 Intervention: For administration of PONV prophylaxis, patients will be randomized into two groups depending upon a computer generated randomized sheet. Group A will receive 8mg of dexamethasone i.v. after anaesthesia induction and 4 mg of ondansetron i.v. 30 minutes prior to the end of surgery. Patients in Group B will be administered 2 mg of midazolam i.v. 30 minutes prior to the end of surgery.

Monitoring and assessment: Patients will be monitored 24 hours post operatively. Any complaints of nausea and/vomiting will be noted and rescue antiemetic will be administered as per the guidelines

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years of age
* Patients belonging to ASA-PS (American society of anesthesiologists Physical status) 1 or 2
* Patients with 2 or more risk factors for developing PONV undergoing laparoscopic surgeries

Exclusion Criteria:

* Anticipated difficult airway
* Obesity (body mass index >30 kg.m2),
* Pregnancy
* Patients with ASA - PS more than 2
* Consumption of an agent with anti-emetic properties within 24 h prior to commencement of the study.
* Known hypersensitivity to midazolam, ondansetron or dexamethasone
* Patients not giving consent.
* Patients with psychiatric illness or mental retardation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea vomiting | 24 hours
  the incidence of postoperative nausea and/or vomiting within first 24 hours postoperatively

SECONDARY OUTCOMES:
Rescue antiemetic | 24 hours
  The amount of antiemetic used within the first 24 hours.
Time to achieve PADSS>9 | 1 hour
  Time taken to achieve a Post anaesthesia discharge score of ≥9
Incidence of PON, POV, PONV at 2 hours and PON and POV at 24 | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kelika Prakash, DM, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India